CLINICAL TRIAL: NCT03129295
Title: A Randomized, Double-Blind, Placebo-Controlled, MultiCenter Study of the Efficacy and Safety of MPC-SHRC for the Relief of Symptoms Associated With Uncomplicated Urinary Tract Infections
Brief Title: Phase II Proof of Concept Study in Uncomplicated UTI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mission Pharmacal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MPC-SHRC-002
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MPC-SHRC (Experimental): oral tablet four times a day for 3 days
  Interventions: Drug: MPC-SHRC
- Placebo (Placebo Comparator): oral tablet four times a day for 3 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: MPC-SHRC — Oral tablet four times a day for 3 days
  Arms: MPC-SHRC
Drug: Placebo Oral Tablet — Oral tablet four times a day for 3 days
  Arms: Placebo

SUMMARY:
A study of the efficacy and safety of MPC-SHRC for the relief of symptoms associated with uncomplicated urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, nonlactating woman with moderate to severe symptoms of urinary tract infection
* On adequate birth control
* Normal ECG

Exclusion Criteria:

* Participated in any other trial within 30 days of visit 1
* Known or suspected allergy to investigational drug
* Narrow angle glaucoma
* Recovering from chicken pox or flu-like symptoms
* History of peptic ulcer, gastrointestinal bleeding, gastrointestinal surgery, or gastrointestinal dysfunction which could interfere with drug absorption
* Taken any drugs for within past 24 hours for symptoms associated with uncomplicated urinary tract infections
* Currently taking prohibited drugs
* Taken an antibiotic within 7 days of Visit 1
* Are ineligible to receive an antibiotic
* History of urinary retention
* History of interstitial cystitis
* History of impaired renal function
* History of impaired hepatic function
* Diagnosis or suspicion of complicated urinary tract infection or systemic infection
* History of substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on assessment instrument | 6 hours after the first dose of study drug
  Patient reported outcome

SECONDARY OUTCOMES:
Change from baseline on assessment instruments | Three hour intervals after first dose of study drug
  Patient reported outcome
Change from baseline on Pain Scale | Three hour intervals after first dose of study drug
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E. Hurley, MD, Study Director — Hurley Consulting Associates Ltd.
Locations (4):
- United States (4):
  - First Urology PSC, Jeffersonville, Indiana
  - Beyer Research, Kalamazoo, Michigan
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey

IPD SHARING:
Plan to Share IPD: No